CLINICAL TRIAL: NCT01260831
Title: Evaluating Processes of Care & the Outcomes of Children in Hospital (EPOCH): a Cluster Randomized Trial of the Bedside Paediatric Early Warning System
Brief Title: Evaluating Processes of Care & the Outcomes of Children in Hospital (EPOCH)
Acronym: EPOCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Christopher Parshuram, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1000018562
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Critically Ill Children
Keywords: BedsidePEWS; Intensive Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Hospitals (Experimental): hospitals randomized to implement bedsidePEWS documentation system (vital sign assessment record)
  Interventions: Other: Implementation of Bedside Paediatric Early Warning System
- Control Hospitals (Active Comparator): hospitals randomized to continue with their pre existing documentation system (vital sign assessment record)
  Interventions: Other: Hospital Standard of Care

INTERVENTIONS:
Other: Implementation of Bedside Paediatric Early Warning System — The Bedside Paediatric Early Warning System (Bedside PEWS) is a documentation-based system of care that will replace existing documentation systems for vital signs in inpatient ward areas in hospitals randomized to implement Bedside-PEWS. Frontline staff education within each hospital will occur over a period of three months preceding a 5 week run-in implementation phase, which will be followed by hospital-wide implementation. The Bedside-PEWS documentation record will become the primary method of documentation for vital signs and related data.
  Arms: Intervention Hospitals
Other: Hospital Standard of Care — Hospitals randomized to standard care will continue with established methods of care. This will include the use of calling criteria and/or the expert model to identify children at risk. As in intervention hospitals, existing MET-RRT practices, established staffing and documentation practices will continue.
  Arms: Control Hospitals

SUMMARY:
The purpose of this study is to evaluate the impact of Bedside Paediatric Early Warning System (Bedside-PEWS) on early identification of children at risk for near and actual cardiopulmonary arrest, hospital mortality, processes of care and PICU resource utilization.

DETAILED DESCRIPTION:
The Bedside Paediatric Early Warning System (Bedside PEWS) is a scientifically developed documentation-based system of care designed to identify children who are clinically deteriorating while admitted to hospital inpatient wards. It was developed and validated by the applicants. The investigators have preliminary data demonstrating that the Bedside PEWS addresses multiple factors (communication, hierarchy, secondary review) contributing to delayed treatment of children at risk. In our pilot study of implementation at a single site the investigators showed statistically significant reductions in late transfers, 'stat' calls, decreased apprehension when nurses called physicians to review patients, and improved communication. Our preliminary data show that the Bedside PEWS score is superior to other methods being used to identify children at risk for impending cardiopulmonary arrest. A 2-year cluster-randomized trial will evaluate the impact of Bedside PEWS on clinical outcomes, processes of care and resource utilization in 22 paediatric hospitals.

ELIGIBILITY:
Inclusion Criteria:

For Hospitals:

* provide care for more than 200 inpatient admissions aged <18 years and >37 weeks gestational age in eligible inpatient wards each year
* have specialised paediatric physicians (including paediatricians, paediatric surgeons, other paediatric sub-specialists) and, one or more intensive care unit (PICU) that provides care for children. A PICU is a designated, staffed area for prolonged mechanical ventilation, invasive monitoring and circulatory support for children- including but not limited to neonates. Other areas designated for patients of increased acuity, such as 'constant observation' or 'high dependency' or 'step-down' units will be regarded as part of the PICU where the PICU staff physicians are wholly or jointly responsible for the care of children in these areas (can write orders in the chart).
* may or may not have a MET-RRT for children. A MET-RRT is defined as an identified team of one or more trained healthcare professionals who report to an on service PICU physician, and perform urgent consultations on hospital inpatients.

For inpatient wards:

* areas where care is provided to patients who are admitted to the hospital, other than PICU, operating rooms, and other designated areas where anaesthetist-supervised procedures are performed. All eligible inpatient wards will participate in the study.

For patients:

Within eligible hospitals we will study patients older than 37 weeks gestational age and less than 18 years who are admitted to eligible inpatient wards, who receive care in an eligible inpatient area during the study.

Exclusion Criteria:

For hospitals:

* have plans to introduce a new 'medical emergency team' during the study, and where a severity of illness score (Brighton, Cardiff, PEWS, Bedside PEWS or other unpublished score) is used in ward areas
* hospitals where randomization is not deemed acceptable. These exclusion criteria ensure that major system changes including introduction of MET-RRT, new documentation systems, physician staffing, and hospital capacity will not bias results.

For patients:

* those who are less than 37 weeks gestational age throughout their hospitalization
* are cared for exclusively in an NICU
* children who are admitted directly to a PICU and die before PICU discharge and thus have not received care in an eligible inpatient ward

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144539 (Actual)
Dates: Start 2011-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
All Cause Hospital Mortality (Intervention Phase) | for 52 weeks starting at Week 31
  All cause hospital mortality includes all deaths of eligible inpatients who were cared for in an eligible inpatient ward and will be prospectively assessed for 52 weeks following the 5-week run in period at intervention hospitals.
  The following sub-group analyses will be performed: [1] Hospital size. Hospitals with >200 eligible inpatient ward beds will be one group and those with <200 eligible inpatient ward beds the other. [2] Hospitals with and without medical emergency teams. [3] Hospitals with ECMO for children. [4] patients with urgent PICU admission initiated in an inpatient ward.

SECONDARY OUTCOMES:
Number of Significant Clinical Deterioration Events | for 26 weeks starting at Week 0 (baseline) and for 52 weeks starting at week 31 (intervention)
  This will be defined as the provision of significant respiratory or circulatory therapies or cardiopulmonary resuscitation in the 12 hours before transfer from inpatient ward, or death without DNR order in an inpatient ward.
  The following sub-group analyses will be performed: [1] Hospital size. Hospitals with >200 eligible inpatient ward beds will be one group and those with <200 eligible inpatient ward beds the other. [2] Hospitals with and without medical emergency teams. [3] Hospitals with ECMO for children. [4] patients with urgent PICU admission initiated in an inpatient ward.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Parshuram, MD, Principal Investigator — The Hospital for Sick Children; Patricia Parkin, Study Chair — The Hospital for Sick Children; James Hutchison, Study Chair — The Hospital for Sick Children; Catherine Farrell, Study Chair — Sainte Justine's Hospital; Martin Gray, Study Chair — St. George's Health Care NHS Trust; Ronald Gottesman, Study Chair — Montreal Children's Hospital of the MUHC; Mark Helfaer, Study Chair — Children's Hospital of Philadelphia; Elizabeth Hunt, Study Chair — Johns Hopkins University; Ari Joffe, Study Chair — Stollery Children's Hospital; Jacques LaCroix, Study Chair — Sainte Justine's Hospital; Vinay Nadkarni, Study Chair — Children's Hospital of Philadelphia; David Wensley, Study Chair — Provincial Health Services Authority British Columbia; Andrew Willan, Study Chair — The Hospital for Sick Children, Research Institute
Locations (22):
- HUDERF: Queen Fabiola Children's University Hospital, Brussels, Belgium
- Canada (11):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - Victoria General Hospital, Victoria, British Columbia
  - Saint John Regional Hospital, Saint John, New Brunswick
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital, Hamilton, Ontario
  - London Health Sciences Center University Hospital, London, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Centre hospitalier universitaire Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - Centre hospitalier universitaire de Québec (CHUQ), Québec
- Ireland (2):
  - Children's University Hospital, Dublin
  - Our Lady's Children's Hospital, Dublin
- Bambino Gesù Children's Hospital, Rome, Italy
- Erasmus MC-Sophia, Rotterdam, Netherlands
- Starship Children's Health, Auckland, New Zealand
- United Kingdom (5):
  - Barts Health - The London NHS Trust, London
  - Kings College Hospital, London
  - Royal Brompton Hospital, London
  - St. George's Hospital, London
  - St. Mary's Hospital - Imperial College Healthcare, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gawronski O, Parshuram CS, Cecchetti C, Tiozzo E, Szadkowski L, Ciofi Degli Atti ML, Dryden-Palmer K, Dall'Oglio I, Raponi M, Joffe AR, Tomlinson G. Evaluating associations between patient-to-nurse ratios and mortality, process of care events and vital sign documentation on paediatric wards: a secondary analysis of data from the EPOCH cluster-randomised trial. BMJ Open. 2024 Jul 4;14(7):e081645. doi: 10.1136/bmjopen-2023-081645. PMID 38964797
- [Derived] Parshuram CS, Dryden-Palmer K, Farrell C, Gottesman R, Gray M, Hutchison JS, Helfaer M, Hunt EA, Joffe AR, Lacroix J, Moga MA, Nadkarni V, Ninis N, Parkin PC, Wensley D, Willan AR, Tomlinson GA; Canadian Critical Care Trials Group and the EPOCH Investigators. Effect of a Pediatric Early Warning System on All-Cause Mortality in Hospitalized Pediatric Patients: The EPOCH Randomized Clinical Trial. JAMA. 2018 Mar 13;319(10):1002-1012. doi: 10.1001/jama.2018.0948. PMID 29486493
- [Derived] Parshuram CS, Dryden-Palmer K, Farrell C, Gottesman R, Gray M, Hutchison JS, Helfaer M, Hunt E, Joffe A, Lacroix J, Nadkarni V, Parkin P, Wensley D, Willan AR; Canadian Critical Care Trials Group. Evaluating processes of care and outcomes of children in hospital (EPOCH): study protocol for a randomized controlled trial. Trials. 2015 Jun 2;16:245. doi: 10.1186/s13063-015-0712-3. PMID 26033094